CLINICAL TRIAL: NCT05117060
Title: A Phase 2 Trial to Evaluate the Efficacy and Safety of Orally Administered LEO 152020 Tablets Compared With Placebo Tablets for up to 16 Weeks of Treatment in Adults With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Safety of LEO 152020 Tablets for the Treatment of Adults With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LP0190-1488; 2020-004561-39 (EudraCT Number); U1111-1281-1895 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-11-08; First posted 2021-11-11 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The outcome assessor is considered to be the person/people who will assess the outcome of the data/study and will in this study therefore be the sponsor.
  To ensure masking across the interventions, each dose of treatment in the LEO 152020 tablet - Dose regimen 2 and LEO 152020 tablet - Dose regimen 3 arms will consist of a combination of LEO 152020 and LEO 152020 placebo tablets. In these arms, placebo will be used as a masking aid and is therefore considered neither a control nor an intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LEO 152020 tablet - Dose regimen 1 (Experimental): Participants will be asked to take tablets from Week 0 to Week 16 (end of treatment).
  Interventions: Drug: LEO 152020 tablet
- LEO 152020 tablet - Dose regimen 2 (Experimental): Participants will be asked to take tablets from Week 0 to Week 16 (end of treatment).
  Interventions: Drug: LEO 152020 tablet; Drug: LEO 152020 placebo tablet
- LEO 152020 tablet - Dose regimen 3 (Experimental): Participants will be asked to take tablets from Week 0 to Week 16 (end of treatment).
  Interventions: Drug: LEO 152020 tablet; Drug: LEO 152020 placebo tablet
- LEO 152020 placebo tablet (Placebo Comparator): Participants will be asked to take tablets from Week 0 to Week 16 (end of treatment).
  Interventions: Drug: LEO 152020 placebo tablet

INTERVENTIONS:
Drug: LEO 152020 tablet — LEO 152020 is a small drug molecule which can bind to the histamine 4 receptor (H4R) and prevent histamine from binding to the receptor. LEO 152020 is a tablet for oral administration.
  Arms: LEO 152020 tablet - Dose regimen 1; LEO 152020 tablet - Dose regimen 2; LEO 152020 tablet - Dose regimen 3
Drug: LEO 152020 placebo tablet — LEO 152020 placebo tablet contains the same excipients in the same concentration as LEO 152020 tablet, except that it does not contain the medical ingredient LEO 152020. LEO 152020 placebo is a tablet for oral administration.
  Arms: LEO 152020 placebo tablet; LEO 152020 tablet - Dose regimen 2; LEO 152020 tablet - Dose regimen 3

SUMMARY:
This is an up to 22-week clinical study in adult participants with moderate to severe atopic dermatitis (AD).

The purpose of the study is to test a new tablet (LEO 152020) to see if it improves AD and what the side effects are when compared with a placebo tablet with no medical ingredient.

During the study, there will be a 16-week treatment period during which the participants will be asked to take the tablets. The participants will regularly visit the clinic for tests and the study doctor will evaluate their AD. The participants will also be asked to answer questions about their AD symptoms, itch, sleep, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 18 years or older at screening.
* Diagnosis of chronic atopic dermatitis (AD).
* History of AD ≥1 year prior to baseline.
* Recent (within 6 months prior to baseline) documented history of inadequate response to topical AD treatments or subject for whom topical AD treatments are medically inadvisable.
* 7.1≤ Eczema Area and Severity Index (EASI) ≤50 at baseline.
* Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) score ≥3 at baseline.

Exclusion Criteria:

* Previous treatment with an oral histidine 4 receptor (H4R) antagonist (including LEO 152020) within 6 months prior to baseline.
* Previous treatment with 3 or more systemic AD treatments prior to screening.
* Women who are pregnant, intend to become pregnant, or are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (43):
- United States (6):
  - LEO Pharma Investigational Site, Beverly Hills, California
  - LEO Pharma Investigational Site, Los Angeles, California
  - LEO Pharma Investigational Site, San Diego, California
  - LEO Pharma Investigational Site, Cincinnati, Ohio
  - LEO Pharma Investigational Site, Murfreesboro, Tennessee
  - LEO Pharma Investigational Site, Frisco, Texas
- Australia (6):
  - LEO Pharma Investigational Site, Darlinghurst, New South Wales
  - LEO Pharma Investigational Site, Kogarah, New South Wales
  - LEO Pharma Investigational Site, Sydney, New South Wales
  - LEO Pharma Investigational Site, Woolloongabba, Queensland
  - LEO Pharma Investigational Site, Carlton, Victoria
  - LEO Pharma Investigational Site, Clayton, Victoria
- Canada (7):
  - LEO Pharma Investigational Site, Calgary, Alberta
  - LEO Pharma Investigational Site, Edmonton, Alberta
  - LEO Pharma Investigational Site, Markham, Ontario
  - LEO Pharma Investigational Site, Mississauga, Ontario
  - LEO Pharma Investigational Site, Niagara Falls, Ontario
  - LEO Pharma Investigational site, Québec, Quebec
  - LEO Pharma Investigational Site, Saint-Jérôme, Quebec
- Czechia (5):
  - LEO Pharma Investigational Site, Karlovy Vary
  - LEO Pharma Investigational Site, Kutná Hora
  - LEO Pharma Investigational Site, Nový Jičín
  - LEO Pharma Investigational Site, Ostrava-Poruba
  - LEO Pharma Investigational Site, Prague
- Germany (5):
  - LEO Pharma Investigational Site, Bad Bentheim
  - LEO Pharma Investigational Site, Berlin
  - LEO Pharma Investigational Site, Hanover
  - LEO Pharma Investigational Site, Magdeburg
  - LEO Pharma Investigational Site, Merzig
- Japan (6):
  - LEO Pharma Investigational Site, Fukuoka, Fukuoka
  - LEO Pharma Investigational Site, Fukutsu-shi, Fukuoka
  - LEO Pharma Investigational Site, Kumamoto, Kumamoto
  - LEO Pharma Investigational Site, Takatsuki-shi, Osaka
  - LEO Pharma Investigational Site, Koto-ku, Tokyo
  - LEO Pharma Investigational Site, Minato-ku, Tokyo
- Poland (5):
  - LEO Pharma Investigational Site, Krakow
  - LEO Pharma Investigational Site, Lodz
  - LEO Pharma Investigational Site, Lublin
  - LEO Pharma Investigational Site, Mikołów
  - LEO Pharma Investigational Site, Wroclaw
- Spain (3):
  - LEO Pharma Investigational Site, Córdoba
  - LEO Pharma Investigational Site, Madrid
  - LEO Pharma Investigational Site, Pontevedra

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Access Criteria: De-identified Individual Participant Data can be made available to researchers and is subject to approved scientifically sound research proposal and signed data-sharing agreement.
URL: http://leopharmatrials.com/for-professionals

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 45 sites that screened subjects in 8 countries (Australia, Canada, Czech Republic (Czechia), Germany, Japan, Poland, Spain and the United States).
Pre-assignment Details: 285 subjects were screened and 216 were randomized in a 4:3:3:4 ratio into the 4 treatment groups.
Groups:
- LEO 152020 - Dosing Regimen 1 (Higher Dose): Subjects administered themselves daily for 16 weeks a fixed treatment of LEO 152020 - higher dose. Film coated tablets, administered orally.
- LEO 152020 - Dosing Regimen 2 (Middle Dose): Subjects administered themselves daily for 16 weeks a fixed treatment of LEO 152020 - middle dose. Film coated tablets, administered orally.
- LEO 152020 - Dosing Regimen 3 (Lower Dose): Subjects administered themselves daily for 16 weeks a fixed treatment of LEO 152020 and LEO 152020 placebo - lower dose. Film coated tablets, administered orally.
- LEO 152020 - Placebo: Subjects administered themselves daily for 16 weeks a fixed treatment of LEO 152020 placebo. Film coated tablets, administered orally.
Period: Overall Study
Arm/Group | LEO 152020 - Dosing Regimen 1 (Higher Dose) | LEO 152020 - Dosing Regimen 2 (Middle Dose) | LEO 152020 - Dosing Regimen 3 (Lower Dose) | LEO 152020 - Placebo
Started | 61 | 45 | 49 | 61
Completed | 44 | 29 | 33 | 46
Not Completed | 17 | 16 | 16 | 15
Not completed — Adverse Event | 3 | 5 | 6 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 4 | 5 | 2 | 6
Not completed — Withdrawal by Subject | 8 | 5 | 5 | 6
Not completed — Other | 2 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 152020 - Dosing Regimen 1 (Higher Dose) | LEO 152020 - Dosing Regimen 2 (Middle Dose) | LEO 152020 - Dosing Regimen 3 (Lower Dose) | LEO 152020 - Placebo | Total
Number analyzed (Participants) | 61 | 45 | 49 | 61 | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2 | 0 | 4
  Between 18 and 65 years | 59 | 40 | 46 | 59 | 204
  >=65 years | 2 | 3 | 1 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (13.3) | 35.2 (15.0) | 35.2 (13.5) | 33.4 (12.9) | 35.0 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 21 | 30 | 35 | 118
  Male | 29 | 24 | 19 | 26 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 17 | 9 | 15 | 14 | 55
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 2 | 2 | 14
  White | 36 | 33 | 30 | 45 | 144
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 1 | 6 | 4 | 14
  Canada | 14 | 6 | 8 | 6 | 34
  Czechia | 5 | 7 | 4 | 12 | 28
  Germany | 8 | 9 | 2 | 8 | 27
  Japan | 10 | 7 | 9 | 10 | 36
  Poland | 12 | 11 | 11 | 14 | 48
  Spain | 2 | 0 | 1 | 1 | 4
  United States | 7 | 4 | 8 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in EASI From Baseline to Week 16
Description: The Eczema Area and Severity Index (EASI) is a validated measure used in clinical trials to evaluate the extent and severity of atopic dermatitis. EASI is a composite score ranging from 0 to 72 with higher scores indicating a more extensive or severe condition.
Time Frame: Week 0 to Week 16
Population: FAS, full analysis set.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LEO 152020 - Dosing Regimen 1 (Higher Dose) | LEO 152020 - Dosing Regimen 2 (Middle Dose) | LEO 152020 - Dosing Regimen 3 (Lower Dose) | LEO 152020 - Placebo
Number analyzed (Participants) | 61 | 45 | 49 | 61
score on a scale | -9.99 [-12.85 to -7.13] | -8.83 [-12.63 to -5.04] | -8.87 [-12.47 to -5.28] | -9.11 [-11.88 to -6.35]

2. Secondary Outcome: Number of Adverse Events From Baseline to Week 16+3 Days Per Subject
Description: Only treatment-emergent adverse events will be reported for this outcome measure. An adverse event will be considered treatment emergent if occurring after the first dose of treatment (Week 0) and up until 3 days after the last dose of treatment (Week 16+3 days for a participant completing the 16-week treatment period).
Time Frame: Week 0 to Week 16+3 days
Population: SAF, safety analysis set
Measure: Number; unit: events
Arm/Group | LEO 152020 - Dosing Regimen 1 (Higher Dose) | LEO 152020 - Dosing Regimen 2 (Middle Dose) | LEO 152020 - Dosing Regimen 3 (Lower Dose) | LEO 152020 - Placebo
Number analyzed (Participants) | 44 | 31 | 33 | 38
events | 109 | 67 | 80 | 75

ADVERSE EVENTS:
Time Frame: Week 0 to Week 16+3 days
Arm/Group | LEO 152020 - Dosing Regimen 1 (Higher Dose) | LEO 152020 - Dosing Regimen 2 (Middle Dose) | LEO 152020 - Dosing Regimen 3 (Lower Dose) | LEO 152020 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/45 | 0/49 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 2/45 | 1/49 | 0/61
Other Adverse Events (participants affected / at risk) | 29/61 | 24/45 | 23/49 | 24/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 152020 - Dosing Regimen 1 (Higher Dose) (N=61) | LEO 152020 - Dosing Regimen 2 (Middle Dose) (N=45) | LEO 152020 - Dosing Regimen 3 (Lower Dose) (N=49) | LEO 152020 - Placebo (N=61)
Eczema herpeticum (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 152020 - Dosing Regimen 1 (Higher Dose) (N=61) | LEO 152020 - Dosing Regimen 2 (Middle Dose) (N=45) | LEO 152020 - Dosing Regimen 3 (Lower Dose) (N=49) | LEO 152020 - Placebo (N=61)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 2 (2) | 5 (5) | 1 (1)
COVID-19 (Infections and infestations) | 6 (6) | 6 (6) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6) | 4 (6) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 2 (3) | 7 (7)
Electrocardiogram QT prolonged (Investigations) | 1 (2) | 3 (3) | 6 (10) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (6)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 10 (14) | 11 (15) | 7 (8) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor seeks publication of all clinical trials in peer-reviewed journals within 12 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by the sponsor within these 12 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT05117060/Prot_SAP_000.pdf